CLINICAL TRIAL: NCT07385495
Title: Analysis of the Expression Profiles of Inflammation-regulating microRNAs in Serum and Tear Samples From Subjects With Allergic Conjunctivitis.
Brief Title: OJO-miR: microRNA Expression in Allergic Conjunctivitis.
Acronym: OJO-miR
Status: Active, not recruiting | Type: Observational
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Principal Investigator, María C. Jiménez Martínez, Head of the Immunology Department, Research Unit, Instituto de Oftalmología Fundación Conde de Valenciana
Other Study IDs: CEI-2025/09/05; Research Committee (Other: CI-069-2025); Biosecurity Committee (Other: CB-069-2025)
Record Dates: First submitted 2026-01-22; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Conjunctivitis, Allergic
Keywords: microRNA; Tears; Serum; Ocular Surface; inflammation
MeSH Terms: conditions — Conjunctivitis, Allergic; Lacerations; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood: Samples are collected following the Institute's Immunology Department manual after verifying informed consent. Personnel must use hand hygiene, masks, and gloves. Venous blood is obtained by venipuncture in Vacutainer tubes with separator gel. Serum is separated by centrifugation and stored at -20°C.
  Tears: Collected according to Santacruz et al. (2015). Personnel must use hand hygiene, gloves, and masks. 20 µL of sterile saline is instilled into each eye. Tear film is collected from the lower lateral meniscus using borosilicate capillaries. Samples are stored in microtubes at -20°C.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with Allergic Conjunctivitis: Subjects aged 5 to 30 years with a confirmed clinical diagnosis of allergic conjunctivitis (Seasonal, Perennial, or Vernal Keratoconjunctivitis). Participants must present active symptomatology and positive skin prick tests corresponding to the allergic condition.
- Healthy Controls: Clinically healthy subjects aged 5 to 30 years with a normal ocular surface evaluation. Participants must have no personal history of allergic diseases (ocular or systemic), no active ocular infection, and no chronic-degenerative or autoimmune diseases.

SUMMARY:
Allergic conjunctivitis (AC) causes inflammation of the conjunctiva in response to environmental allergens, affecting a significant percentage of the world population and reducing quality of life. The pathophysiology is poorly understood, lacking effective treatments. MicroRNAs have potential for diagnosing and characterizing inflammatory diseases. This study aims to compare the expression profiles of inflammation-regulating microRNAs (miR-19, miR-23, miR-125b, miR-146a, and miR-155) in serum and tear samples from subjects with AC and healthy subjects to identify biomarkers and therapeutic targets.

DETAILED DESCRIPTION:
Allergic conjunctivitis (AC) is an inflammatory disorder of the conjunctiva triggered by exposure to environmental allergens. This ocular condition affects a significant proportion of the global population, leading to a reduction in quality of life and, in some cases, visual impairment. The pathophysiology of AC remains poorly understood, and effective targeted therapies are limited. MicroRNAs have emerged as promising tools for the diagnosis and characterization of inflammatory diseases such as asthma and rhinitis; however, studies evaluating microRNA involvement in allergic conjunctivitis are scarce. Therefore, identifying microRNAs that are differentially regulated in AC is essential to better understand disease pathogenesis and to explore potential biomarkers and therapeutic targets.

This study aims to determine whether differences exist in the expression profiles of inflammation-regulatory microRNAs between subjects with allergic conjunctivitis and healthy controls. The working hypothesis is that subjects with allergic conjunctivitis exhibit differential expression of inflammation-related microRNAs compared with healthy individuals.

An observational cross-sectional study will be conducted including subjects aged 5 to 30 years with a clinical diagnosis of allergic conjunctivitis, as well as age-matched healthy controls. Tear samples and peripheral blood samples for serum isolation will be collected from all participants. Total RNA will be extracted from both sample types, and the expression of miR-19, miR-23, miR-125b, miR-146a, and miR-155 will be quantified using quantitative real-time polymerase chain reaction (qRT-PCR). Relative expression levels (fold change) will be calculated in the allergic conjunctivitis group and compared with those observed in healthy controls to identify microRNAs specifically associated with the disease. Receiver operating characteristic (ROC) curve analysis will be performed to evaluate the potential of the studied microRNAs as diagnostic biomarkers.

ELIGIBILITY:
Inclusion Criteria

* Subjects with Allergic Conjunctivitis:
* Age between 5 and 30 years.
* Clinical diagnosis of allergic conjunctivitis.
* Presence of active ocular symptoms at the time of sample collection.
* Positive skin prick test.
* Written informed consent signed by the participant or parent/legal guardian, -with assent when applicable.

Healthy Controls:

* Age between 5 and 30 years.
* Clinically healthy subjects with a normal ocular surface.
* No evidence of active ocular disease.
* Written informed consent signed by the participant or parent/legal guardian, with assent when applicable.

Exclusion Criteria

* Subjects with Allergic Conjunctivitis:
* History of infectious disease within 2 months prior to sample collection.
* Presence of active systemic allergic diseases (e.g., asthma, active dermatitis).
* Chronic degenerative or autoimmune diseases.
* Use of topical immunosuppressive treatment within 2 months prior to sample collection.
* Use of systemic immunosuppressive therapy.

Healthy Controls:

-History of infectious disease within 2 months prior to sample collection.

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population will include subjects aged 5 to 30 years with a clinical diagnosis of allergic conjunctivitis, as well as age-matched healthy controls. Participants will be recruited from a specialized ophthalmology center. Subjects with allergic conjunctivitis must present active ocular symptoms at the time of enrollment, while healthy controls must have a clinically normal ocular surface and no history of active ocular disease. All participants or their legal guardians will provide written informed consent, with assent obtained from minors when applicable.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-01-05 (Estimated); Study Completion 2027-07-05 (Estimated)

PRIMARY OUTCOMES:
Expression of inflammation-regulatory microRNAs in tear samples | Baseline
  Relative expression (fold change) of miR-19, miR-23, miR-125b, miR-146a, and miR-155 in tear samples measured by quantitative real-time polymerase chain reaction (qRT-PCR) and calculated using the 2^-ΔΔCT method.
Expression of inflammation-regulatory microRNAs in serum samples | Baseline
  Relative expression (fold change) of miR-19, miR-23, miR-125b, miR-146a, and miR-155 in serum samples measured by quantitative real-time polymerase chain reaction (qRT-PCR) and calculated using the 2^-ΔΔCT method.

SECONDARY OUTCOMES:
Diagnostic performance of candidate microRNAs | Baseline
  Evaluation of the diagnostic potential of miR-19, miR-23, miR-125b, miR-146a, and miR-155 through receiver operating characteristic (ROC) curve analysis, including area under the curve (AUC).

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmología FAP Conde de Valenciana, IAP Sede Centro, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No